CLINICAL TRIAL: NCT05274464
Title: A Recurrence Nomogram to Guide Surveillance Strategies After the Resection of Hepatoid Adenocarcinoma of the Stomach: a China Hepatoid Adenocarcinoma of the Stomach Study Group Database Study
Brief Title: A Recurrence Nomogram for Hepatoid Adenocarcinoma of the Stomach
Status: Completed | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University
Other Study IDs: HAS-GC-01
Record Dates: First submitted 2022-03-02; First posted 2022-03-10 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Gastric Cancer
Keywords: Reurrence-free survival; Nomogram
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to develop a nomogram to predict postoperative recurrence of HAS and guide individually tailored surveillance strategies.

DETAILED DESCRIPTION:
Patients were included from the China Hepatoid Adenocarcinoma of the Stomach Study Group (China-HASSG) database, which comprises 14 tertiary referral centers. All the patients who had undergone complete resection of a primary HAS between April 2004 and December 2019 were included. First, univariate analysis was performed in Cox regression to identify the risk factors associated with RFS. Next, variables with P< 0.05 in univariable analysis were included in the multivariable model, and the forward likelihood ratio method was used for analysis to confirm the independent prognostic factors associated with RFS. Finally, based on the results of multivariable analysis, variables that achieved significance at P< 0.05 were selected to formulate a nomogram.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had undergone complete resection of a primary HAS between April 2004 and December 2019

Exclusion Criteria:

* Patients with metastatic disease, patients who had undergone palliative surgery, patients who had died within 30 days, and patients who were lost to follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with primary HAS who had undergone curative-intent resection at 14 institutions in China from 2004 to 2019 were included.
Sampling Method: Non-Probability Sample
Enrollment: 261 (Actual)
Dates: Start 2004-04-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Reurrence-free survival | 3 year
  Reurrence-free survival was defined as the time interval from the date of the operation to the date of first recurrence or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China